CLINICAL TRIAL: NCT04446494
Title: Identification and Preservation of Arm Lymphatics (DEPART) in Axillary Dissection for Breast Cancer to Reduce Arm Lymphedema Events: A Multicenter Randomized Clinical Trial
Brief Title: Identification and Preservation of Arm Lymphatics
Acronym: DEPART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Gaosong Wu, Ph D, MD, Chair, Department of Thyroid and Breast Surgery, Zhongnan Hospital of Wuhan University, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZLYNXM202014
Record Dates: First submitted 2020-06-21; First posted 2020-06-25 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer Related Lymphedema
Keywords: breast cancer; axillary lymph node dissection; lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Axillary dissection with DEPART technique (Experimental): In the experimental group, 1 ml (2.5 mg) indocyanine green (ICG) and methylene blue (MB) was intradermally injected into the internal bicipital sulcus of ipsilateral arm. During axillary dissection, the identified arm sentinel nodes were carefully injected with 0.1 ml methylene blue (MB) using a 1-cc syringe with a 32-gauge needle. MB could then flow from the nodes along several lymphatic channels toward the infraclavicular nodes. Subsequent-echelon nodes and lymphatics were identified. Sentinel lymph nodes (SLNs) were removed after the identification of the arm sentinel nodes and the procedure of MB injection. When patients harbored positive SLNs, axillary lymph node dissection (ALND) was performed subsequently. All discernible arm lymphatics and lymph nodes were preserved, except that gross arm lymph nodes (major axis larger than 10 mm or node firm on palpation) were sent for immediate partial frozen section (pFS) to determine their resection during ALND.
  Interventions: Procedure: Identification and preservation of arm lymphatics (DEPART)
- Standard axillary dissection (No Intervention): In the control group (no intervention), ALND was performed with complete resection of at least Berg's levels I and II. Resection of level III was performed only in cases with gross disease in level II and/or III

INTERVENTIONS:
Procedure: Identification and preservation of arm lymphatics (DEPART) — Indocyanine green was utilized to identify arm sentinel nodes, and 0.1 ml MB was injected into the arm sentinel nodes to reveal the subsequent-echelon nodes and lymphatics. Gross arm lymph nodes were examined by intraoperative partial frozen section and were removed if positive.
  Arms: Axillary dissection with DEPART technique

SUMMARY:
Controversy in axillary reverse mapping in axillary lymph node dissection (ALND) possibly results from incomplete recognition of the arm lymphatic system (ALS) and its compromise to oncological safety. The iDEntification and Preservation of ARm lymphaTics (DEPART) technique facilitates complete identification of ALS; therefore, its use may decrease the occurrence of arm lymphedema. This study aimed to examine the arm lymphedema rate, locoregional recurrence, and feasibility to perform DEPART in ALND.

In the study group, indocyanine green and methylene blue (MB) were utilized to identify arm sentinel nodes, and 0.1 ml MB was injected into the arm sentinel nodes to reveal the subsequent-echelon nodes and lymphatics. Gross arm lymph nodes were examined by intraoperative partial frozen section and were removed if positive. Arm lymphedema, local recurrence, regional recurrence, and distant metastasis were recorded at different follow-up examinations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with T1-3 invasive breast cancer;
* Clinically node-positive breast cancer, defined as positive on preoperative axillary palpation, ultrasound examination, and computed tomography scan with contrast;
* Patients who underwent mastectomy with a positive sentinel lymph node (SLN);
* Patients who underwent breast-conserving surgery containing more than two positive SLNs.

Exclusion Criteria:

* Neoadjuvant chemotherapy;
* Previous history of breast cancer.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of arm lymphedema | Up to 2 years
  A difference in volume between the arms < 10% was defined as lymphedema.

SECONDARY OUTCOMES:
Rate of locoregional recurrence | 5-year estimate reported after a median follow-up of 60 months
  Locoregional recurrence included local recurrence and regional recurrence. Local recurrence was defined as chest wall recurrence of breast cancer, and regional recurrence was defined as the axilla recurrence of breast cancer.
Rate of distant metastasis | 5-year estimate reported after a median follow-up of 60 months
  Cancer cells from breast metastasized to other organs.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yuan Q, Wu G, Xiao SY, Hou J, Ren Y, Wang H, Wang K, Zhang D. Identification and Preservation of Arm Lymphatic System in Axillary Dissection for Breast Cancer to Reduce Arm Lymphedema Events: A Randomized Clinical Trial. Ann Surg Oncol. 2019 Oct;26(11):3446-3454. doi: 10.1245/s10434-019-07569-4. Epub 2019 Jun 25. PMID 31240591